CLINICAL TRIAL: NCT06637176
Title: Laser Speckle Contrast Imaging for Intraoperative Assessment of Anastomotic Perfusion
Brief Title: Examination of the Blood Supply of the Intestine Before Suturing the Ends of the Intestine.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Viborg Regional Hospital (Other); Randers Regional Hospital (Other); Gødstrup Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2314383; Doc.nr.: 2913575 (Registry Identifier: The Medical Scientific Ethics Committees Denmark)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-04

CONDITIONS: Surgical Procedure, Unspecified
Keywords: microcirculation; surgical decision making; colon surgery
MeSH Terms: interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Colon Surgery with Extracorporeal Anastomosis: All individuals over 18 years old undergoing elective colon surgery with the formation of an extracorporeal anastomosis are eligible to participate, regardless of indication, comorbidities, or other conditions.
  Interventions: Device: Laser speckle contrast imaging

INTERVENTIONS:
Device: Laser speckle contrast imaging — LSCI measurements will be taken before and after the formation of the anastomosis, with the surgeon blinded to the measurements to prevent any influence on surgical decision-making. The surgery will be performed as standard-of-care, unaffected by the LSCI measurements.
  Following the surgery, the LSCI images will be presented to the surgeon, who will complete a questionnaire assessing whether the LSCI images, if presented perioperatively, would have influenced their decision regarding the location of the anastomotic site. Additionally, the surgeon will be asked if they consider LSCI to be a useful intraoperative tool in general. The surgical case and the series of LSCI images will also be presented to an independent surgeon, who will answer the same set of questions.
  The LSCI measurements will be correlated with 30-day complication rates, with a specific focus on anastomotic leakage (AL).
  Microcirculation is assessed using LSCI at a wavelength of 785 nm (MoorFLPI-2, Moor Instruments

SUMMARY:
In this non-interventional, multicenter study in the Central Denmark Region, the potential of assessing blood supply during colorectal surgery will be explored using a recognized and reliable laser technique called Laser Speckle Contrast Imaging. The study aims to evaluate whether surgeons find this tool valuable in the decision-making process regarding where to perform the anastomosis during the operation.

DETAILED DESCRIPTION:
Anastomotic leakage (AL) is among the most severe and feared postoperative complications of colorectal surgery as it is directly associated with an increase in mortality and morbidity. AL increases risk of local recurrence, decreases the 5-year survival rate, and impairs the patient's quality of life. Despite improvements in the surgical technique, AL continues to occur with high frequency. The cause of AL is considered multifactorial and several factors have shown association with increased risk of AL, although the complete pathogenesis is still unclear; It is recognized that one of the most important risk factors is inadequate blood supply to the anastomotic site, since optimal perfusion is essential for the healing of the anastomosis.

Currently, the assessment of the perfusion at the anastomotic site is based on a subjective clinical estimate by the surgeon (e.g., palpable pulsation of the arteries in the mesenterium, normal color of the intestine, bleeding from the surgical edges, and/or pulsatile bleeding from marginal arteries). However, these assessments are shown to lack objectivity, quantifiability, and predictive accuracy - even experienced surgeons underestimate the risk of AL.

Preventing AL is crucial for improving the outcomes of colorectal surgery. Studies have shown that understanding the state of microcirculation can help reduce the rate of AL. Therefore, having an accurate evaluation of local intestinal microcirculation is the first step in aiding surgeons to make informed decisions on the optimal anastomotic side.

Laser Speckle Contrast Imaging (LSCI) is a dye-free non-contact, non-invasive image-based method, capable of quantitative estimation of the local intestinal perfusion. Further, it allows for time-independent repeated measurements. LSCI uses laser light to generate a speckle pattern: When an object is in motion or contains moving particles such as blood cells, the interference between beams is affected, leading to variations in the phases and the creation of a dynamic speckle pattern. Based on the movements of the red blood cells, LSCI can be used to assess the blood flow within the tissue (microcirculation). Thus, LSCI cannot measure absolute flow but rather measures contrast changes and results are expressed as flux in arbitrary laser speckle perfusion units (LSPU), where higher LSPU values correspond to better tissue perfusion. LSCI is validated and used in small animal and human studies of the gastro-intestinal tract but has not yet been thoroughly tested in a true clinical setting.

LSCI has been utilized in various clinical contexts, including the gastrointestinal system, demonstrating ease and safety of use. However, there is only one similar study from 2019 in Japan where measurements were conducted on 8 patients undergoing colon surgery. The limitations of this study include its single-center nature, involvement of only one surgeon, and a lack of description regarding the surgeons' perspectives on LSCI measurements - whether they consider it a useful tool in their intraoperative procedures. Recently, another study has been published employing LSCI to measure the colon intraoperatively. Nevertheless, this study utilizes a newly developed laparoscopic-based LSCI technique, and it compares surgeons' subjective assessments of the technique. The findings indicate a high level of satisfaction, with 67% of surgeons expressing a willingness to make changes during surgery based on the images. Despite numerous clinical studies supporting the feasibility of LSCI, the literature on colon surgery lacks sufficient evidence to generalize the use of open LSCI equipment across all operating rooms as a tool for surgeons, despite its demonstrated potential.

It is hypothesized that LSCI is a method that could help surgeons evaluate and qualify the peri-operative intestinal microcirculation when anastomoses are formed.

The aim of this study is to investigate this hypothesis.

Study objectives:

1. To provide a descriptive analysis of using LSCI during colorectal surgery to assess microcirculation in the intestines before and after anastomosis formation and evaluate the feasibility of the method.
2. To assess the surgeon's subjective perception whether LSCI could be a useful tool to aid their decision-making during surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing any elective colorectal surgery with the potential formation of an extracorporeal anastomosis as part of the surgical procedure are eligible for inclusion, irrespective of the indication for surgery. Patients will be consecutively included, after informed consent.

Exclusion Criteria:

* In this clinical feasibility trial, exclusion criteria apply only in cases where the inclusion criteria are not met or if performing an extracorporeal anastomosis is not feasible during surgery. Otherwise, patients meeting the inclusion criteria will be considered eligible for participation in the trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified and included from the Regional Hospital Gødstrup, Viborg, and Randers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of using LSCI during colorectal surgery | from enrollment to surgery, aroundt 1-2 weeks.
  The operation time and the time required to perform LSCI will be recorded. It is predefined that an acceptable LSCI duration will be a maximum of 5% of the total operation time.
Descriptive analysis of using LSCI during colorectal surgery | from enrollment to surgery, aroundt 1-2 weeks.
  The number of times the sterile field is breached, the nature of each breach, and whether the breach can be rectified will be recorded. An acceptable sterile breach rate is predefined at 95%, and LSCI will only be considered feasible if 100% of the breaches are mendable.
Descriptive analysis of using LSCI during colorectal surgery | from enrollment to surgery, aroundt 1-2 weeks.
  The number of LSCI measurement attempts made for each patient before a successful final measurement is obtained will be recorded. It is predefined that up to two attempts per successful LSCI measurement is considered acceptable.
Descriptive analysis of using LSCI during colorectal surgery | from enrollment to surgery, aroundt 1-2 weeks.
  Surgeons will be asked, through a questionnaire, for their subjective opinion on whether LSCI in any way disturbs or interferes with the standard procedure in an unacceptable manner. It is predefined that LSCI will not be considered disruptive to the surgical procedure if more than 90% of surgeons find it acceptable.

SECONDARY OUTCOMES:
Assess the surgeon's subjective perception whether LSCI could be a useful tool to aid their decision-making during surgery | from enrollment to surgery, aroundt 1-2 weeks.
  By questionnaire, surgeons are asked their subjective opinion on whether LSCI is a useful intraoperative tool. The endpoint is expressed as the percentage of surgeons who subjectively find LSCI will be a useful tool.
Assess the surgeon's subjective perception whether LSCI could be a useful tool to aid their decision-making during surgery | from enrollment to surgery, aroundt 1-2 weeks.
  By questionnaire, surgeons are asked their subjective opinion on whether they would have changed their intestinal resection line or anastomosis site if LSCI measurements were available during the operation. The endpoint is expressed at the percentage of surgeons who would have changed the resection line or anastomotic site if LSCI measurements had been available.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Region hospital Gødstrup, Herning
  - Region Hospital Randers, Randers
  - Region Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No
There are so few patients that Danish GDP data cannot be shared as it cannot be anonymized, which would be in violation of Danish data protection law.

REFERENCES:
- [Background] Heeman W, Calon J, van der Bilt A, Pierie JEN, Pereboom I, van Dam GM, Boerma EC. Dye-free visualisation of intestinal perfusion using laser speckle contrast imaging in laparoscopic surgery: a prospective, observational multi-centre study. Surg Endosc. 2023 Dec;37(12):9139-9146. doi: 10.1007/s00464-023-10493-0. Epub 2023 Oct 9. PMID 37814165
- [Background] Kojima S, Sakamoto T, Nagai Y, Matsui Y, Nambu K, Masamune K. Laser Speckle Contrast Imaging for Intraoperative Quantitative Assessment of Intestinal Blood Perfusion During Colorectal Surgery: A Prospective Pilot Study. Surg Innov. 2019 Jun;26(3):293-301. doi: 10.1177/1553350618823426. Epub 2019 Jan 13. PMID 30638132
- [Background] Paramasivam R, Kristensen NM, Ambrus R, Stavsetra M, Orntoft MB, Madsen AH. Laser speckle contrast imaging for intraoperative assessment of intestinal microcirculation in normo- and hypovolemic circulation in a porcine model. Eur Surg Res. 2023 Dec 7. doi: 10.1159/000535525. Online ahead of print. PMID 38061337